CLINICAL TRIAL: NCT02916615
Title: Diet and Nitric Oxide (DINO): A Study on the Effects of Dietary Nitrate on Blood Pressure in Subjects With Prehypertension
Brief Title: Effects of Nitrate in Vegetables on Blood Pressure in Subjects With Prehypertension
Acronym: DINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jon Lundberg, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DINO1
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Hypertension; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Nitrates; potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High nitrate vegetables (Active Comparator): During 5 weeks subjects receive 100-150 g of a leafy green vegetable (High nitrate vegetables) per day and placebo pills containing 300 mg KCl (2 x 150 mg).
  Interventions: Other: High nitrate vegetables
- Low nitrate vegetables (Placebo Comparator): During 5 weeks subjects receive 100-150 g of tomatoes/sweet pepper (Low nitrate vegetables) per day and placebo pills containing 300 mg KCl (2 x 150 mg).
  Interventions: Other: Low nitrate vegetables
- Low nitrate vegetables + nitrate (Active Comparator): During 5 weeks subjects receive 100-150 g of tomatoes/sweet pepper (Low nitrate vegetables) per day and nitrate pills containing 300 mg KNO3 (2 x 150 mg).
  Interventions: Dietary Supplement: Low nitrate vegetables + nitrate

INTERVENTIONS:
Other: High nitrate vegetables — vegetables naturally high in nitrate
  Arms: High nitrate vegetables
Dietary Supplement: Low nitrate vegetables + nitrate — pill containing KNO3
  Other Names: potassium nitrate (KNO3)
  Arms: Low nitrate vegetables + nitrate
Other: Low nitrate vegetables — vegetables naturally low in nitrate
  Arms: Low nitrate vegetables

SUMMARY:
The purpose of this study is to examine the effect of different vegetables on cardiovascular function in subjects with moderately increased blood pressure. Specifically we are comparing the effects of vegetables with a high natural content of inorganic nitrate with those of vegetables with a low nitrate content.

DETAILED DESCRIPTION:
Recent studies indicate that dietary-derived inorganic nitrate can affect blood pressure in humans by converting into nitric oxide bioactivity. Here we will study if vegetables that naturally contain high amounts of nitrate (green leafy vegetables) can lower blood pressure and whether any effect is attributed to the nitrate anion. High nitrate vegetables are compared with vegetables low in nitrate (e.g. tomatoes, sweet pepper). After a 2 week run in period where all subjects receive vegetables low in nitrate, the participants are randomized to one of three interventions. One third of the patients receive high-nitrate vegetables + a placebo pill (KCl), one third receives low-nitrate vegetables + placebo and the third group receives low-nitrate vegetables + a nitrate pill (KNO3). The nitrate content in the pill is precisely matched to the nitrate content in the high-nitrate vegetable group.

ELIGIBILITY:
Inclusion Criteria:

Age 50-70 years Systolic blood pressure >130 at screening visit 2

Exclusion Criteria:

Systolic blood pressure <120 or >159 mm Hg at screening 2 Systolic blood pressure > 169 mm Hg at screening 1 Chronic kidney disease Chronic rheumatic disease Insulin treated diabetes mellitus Atrial fibrillation Major cardiovascular event within 6 months Inflammatory bowel disease Malignancy, actively treated within 6 months Hepatitis Polycytemia Vera

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Difference in Change in ambulatory Systolic Blood Pressure From Baseline | 5 weeks intervention
  Measure how 24h ambulatory SBP changes over 5 weeks with the different interventions

SECONDARY OUTCOMES:
Difference in Change in ambulatory diastolic Blood Pressure From Baseline | 5 weeks intervention
  Measure how 24h ambulatory DBP changes over 5 weeks with the different interventions
Difference in Change in office diastolic blood pressure (DBP) | Once every week for 5 weeks
  BP is measured during a hospital visit every week during intervention
Difference in Change in flow mediated dilatation (FMD) | 5 weeks intervention
  FMD is measured before and after the interventions
Difference in Change in office Systolic Blood Pressure From Baseline | 5 weeks intervention
  Measure how clinic SBP changes weekly over 5 weeks with the different interventions
Difference in Change in Daytime Ambulatory systolic Blood Pressure From Baseline | 5 weeks intervention
  Measure how 24h ambulatory daytime SBP changes over 5 weeks with the different interventions

CONTACTS AND LOCATIONS:
Overall Officials: Jon Lundberg, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sundqvist ML, Larsen FJ, Carlstrom M, Bottai M, Pernow J, Hellenius ML, Weitzberg E, Lundberg JO. A randomized clinical trial of the effects of leafy green vegetables and inorganic nitrate on blood pressure. Am J Clin Nutr. 2020 Apr 1;111(4):749-756. doi: 10.1093/ajcn/nqaa024. PMID 32091599